CLINICAL TRIAL: NCT01531374
Title: Medtronic CoreValve® Continued Access Study
Brief Title: Safety and Efficacy Continued Access Study of the Medtronic CoreValve® System in the Treatment of Symptomatic Severe Aortic Stenosis in Very High Risk Subjects and High Risk Subjects Who Need Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10037989DOC REV 1C
Record Dates: First submitted 2012-02-03; First posted 2012-02-10 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Severe Aortic Stenosis
Keywords: Valvular Heart Disease; Critical Aortic Stenosis; Severe Aortic Stenosis; Extreme Risk; High Risk; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Extreme Risk: TAVI Iliofemoral (Experimental): Extreme Risk Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI); Iliofemoral Access
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- Extreme Risk: TAVI Non-Iliofemoral (Experimental): Extreme Risk Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI); Non-Iliofemoral Access
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- High Risk: TAVI (Experimental): High Risk Surgical Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of the Medtronic CoreValve® System in the treatment of symptomatic severe aortic stenosis in subjects who have a predicted very high risk and high risk for aortic valve surgery.

ELIGIBILITY:
Inclusion Criteria:

1. High Risk: Subject must have co-morbidities such that one cardiologist and two cardiac surgeons agree that predicted risk of operative mortality is ≥15% (and predicted operative mortality or serious, irreversible morbidity risk of < 50%) at 30 days.

   OR

   Extreme Risk: Subject must have co-morbidities such that one cardiologist and two cardiac surgeons agree that medical factors preclude operation, based on a conclusion that the probability of death or serious morbidity exceeds the probability of meaningful improvement. Specifically, the predicted operative risk of death or serious, irreversible morbidity is ≥ 50% at 30 days.
2. Subject has senile degenerative aortic valve stenosis with:

   * Mean gradient > 40 mmHg, or jet velocity greater than 4.0 m/sec by either resting or dobutamine stress echocardiogram, or simultaneous pressure recordings at cardiac catheterization (either resting or dobutamine stress), AND
   * An initial aortic valve area of ≤ 0.8 cm2 (or aortic valve area index ≤ 0.5 cm2/m2) by resting echocardiogram or simultaneous pressure recordings at cardiac catheterization
3. Subject is symptomatic from his/her aortic valve stenosis, as demonstrated by New York Heart Association (NYHA) Functional Class II or greater.
4. The subject or the subject's legal representative has been informed of the nature of the trial, agrees to its provisions and has provided written informed consent as approved by the IRB of the respective clinical site.
5. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

Exclusion Criteria:

Clinical

1. Evidence of an acute myocardial infarction ≤ 30 days before the intended treatment.
2. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the MCS TAVI procedure including bare metal and drug eluting stents.
3. Blood dyscrasias as defined: leukopenia (WBC < 1000mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy.
4. Untreated clinically significant coronary artery disease requiring revascularization.
5. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
6. Need for emergency surgery for any reason.
7. Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20% as measured by resting echocardiogram.
8. Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
9. End stage renal disease requiring chronic dialysis or creatinine clearance < 20 cc/min.
10. Active GI bleeding that would preclude anticoagulation.
11. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated:

    * Aspirin
    * Heparin (HIT/HITTS) and bivalirudin
    * Nitinol (titanium or nickel)
    * Ticlopidine and clopidogrel
    * Contrast media
12. Ongoing sepsis, including active endocarditis.
13. Subject refuses a blood transfusion.
14. Life expectancy < 12 months due to associated non-cardiac co-morbid conditions.
15. Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent.
16. Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
17. Currently participating in an investigational drug or another device trial.
18. Symptomatic carotid or vertebral artery disease.

    Anatomical
19. High Risk:Native aortic annulus size < 20 mm or > 29 mm per the baseline diagnostic imaging (until 23mm valve enrollment completion/closure in the CoreValve® US Pivotal Trial-High Risk Cohort)

    OR

    Extreme Risk: Native aortic annulus size < 18 mm or > 29 mm per the baseline diagnostic imaging. (High risk and extreme risk upon 23mm valve enrollment completion/closure in the CoreValve® US Pivotal Trial-High Risk Cohort)
20. Pre-existing prosthetic heart valve any position.
21. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation (3-4+)).
22. Moderate to severe (3-4+) or severe (4+) mitral or severe (4+) tricuspid regurgitation.
23. Moderate to severe mitral stenosis.
24. Hypertrophic obstructive cardiomyopathy.
25. Echocardiographic evidence of new or untreated intracardiac mass, thrombus or vegetation.
26. Severe basal septal hypertrophy with an outflow gradient.
27. Aortic root angulation (angle between plane of aortic valve annulus and horizontal plane/vertebrae) > 70° (for femoral and left subclavian/axillary access) and > 30° (for right subclavian/axillary access).
28. Ascending aorta diameter >43 mm if the aortic annulus diameter is 23-29 mm; ascending aortic diameter > 40 mm if the aortic annulus diameter is 20-23 mm; or an ascending aorta diameter > 34 mm if the aortic annulus diameter is 18-20 mm (Extreme Risk only until 23 mm valve enrollment completion/closure in the CoreValve® US Pivotal Trial-High Risk Cohort).
29. Congenital bicuspid or unicuspid valve verified by echocardiography.
30. Sinus of valsalva anatomy that would prevent adequate coronary perfusion.

    Vascular
31. Transarterial access not able to accommodate an 18Fr sheath.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2777 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Adams, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (45):
- United States (45):
  - Banner Good Samaritan, Phoenix, Arizona
  - University of Southern California University Hospital, Los Angeles, California
  - Kaiser Permanente - Los Angeles Medical Center, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington Hospital Center / Georgetown Hospital, Washington D.C., District of Columbia
  - University of Miami Health System / Jackson Memorial Hospital, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Cardiovascular Institute of the South/Terrebonne General, Houma, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Detroit Medical Center Cardiovascular Institute, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Morristown Memorial Hospital, Morristown, New Jersey
  - North Shore University Hospital/ Long Island Jewish Hospital, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University - Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals - Case Medical Center, Cleveland, Ohio
  - The Ohio State University Medical Center - The Richard M. Ross Heart Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pinnacle Health, Harrisburg, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Texas Heart Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital - The Methodist DeBakey Heart & Vascular Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - St. Luke's Medical Center - Aurora Health Care, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Yakubov SJ, Van Mieghem NM, Oh JK, Ito S, Grubb KJ, O'Hair D, Forrest JK, Gada H, Mumtaz M, Deeb GM, Tang GHL, Rovin JD, Jain R, Windecker S, Skelding KA, Kleiman NS, Chetcuti SJ, Dedrick A, Boatman SV, Popma JJ, Reardon MJ. Impact of Transcatheter or Surgical Aortic Valve Performance on 5-Year Outcomes in Patients at >/= Intermediate Risk. J Am Coll Cardiol. 2025 Apr 8;85(13):1419-1430. doi: 10.1016/j.jacc.2025.02.009. Epub 2025 Mar 9. PMID 40175015
- [Derived] Klautz RJM, Rao V, Reardon MJ, Deeb GM, Dagenais F, Moront MG, Little SH, Labrousse L, Patel HJ, Ito S, Li S, Sabik JF 3rd, Oh JK. Examining the typical hemodynamic performance of nearly 3000 modern surgical aortic bioprostheses. Eur J Cardiothorac Surg. 2024 May 3;65(5):ezae122. doi: 10.1093/ejcts/ezae122. PMID 38710669
- [Derived] O'Hair D, Yakubov SJ, Grubb KJ, Oh JK, Ito S, Deeb GM, Van Mieghem NM, Adams DH, Bajwa T, Kleiman NS, Chetcuti S, Sondergaard L, Gada H, Mumtaz M, Heiser J, Merhi WM, Petrossian G, Robinson N, Tang GHL, Rovin JD, Little SH, Jain R, Verdoliva S, Hanson T, Li S, Popma JJ, Reardon MJ. Structural Valve Deterioration After Self-Expanding Transcatheter or Surgical Aortic Valve Implantation in Patients at Intermediate or High Risk. JAMA Cardiol. 2023 Feb 1;8(2):111-119. doi: 10.1001/jamacardio.2022.4627. PMID 36515976
- [Derived] Butala NM, Song Y, Shen C, Cohen DJ, Yeh RW. Effect of intensive versus limited monitoring on clinical trial conduct and outcomes: A randomized trial. Am Heart J. 2022 Jan;243:77-86. doi: 10.1016/j.ahj.2021.09.002. Epub 2021 Sep 14. PMID 34529944
- [Derived] Pineda AM, Kevin Harrison J, Kleiman NS, Reardon MJ, Conte JV, O'Hair DP, Chetcuti SJ, Huang J, Yakubov SJ, Popma JJ, Beohar N. Clinical impact of baseline chronic kidney disease in patients undergoing transcatheter or surgical aortic valve replacement. Catheter Cardiovasc Interv. 2019 Mar 1;93(4):740-748. doi: 10.1002/ccd.27928. Epub 2018 Oct 20. PMID 30341970
- [Derived] Kleiman NS, Maini BJ, Reardon MJ, Conte J, Katz S, Rajagopal V, Kauten J, Hartman A, McKay R, Hagberg R, Huang J, Popma J; CoreValve Investigators. Neurological Events Following Transcatheter Aortic Valve Replacement and Their Predictors: A Report From the CoreValve Trials. Circ Cardiovasc Interv. 2016 Sep;9(9):e003551. doi: 10.1161/CIRCINTERVENTIONS.115.003551. PMID 27601429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 21, 2012 and April 15, 2014, 1658 subjects were enrolled in the Continued Access Extreme Risk Study at 45 centers in the US. Between October 19, 2012 and August 12, 2014, 1119 subjects were enrolled in the High Risk Study at the same 45 US centers.
Groups:
- Extreme Risk: Iliofemoral: Extreme Risk Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI); Iliofemoral Access
  Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- Extreme Risk: Non-Iliofemoral: Extreme Risk Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI); Non-Iliofemoral Access
  Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- High Risk: High Risk Surgical Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
Period: Overall Study
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Started | 1285 | 373 | 1119
Completed | 921 | 231 | 836
Not Completed | 364 | 142 | 283

BASELINE CHARACTERISTICS:
Population: A total of 1658 Extreme Risk subjects were enrolled; 1257 Iliofemoral and 367 Non-Iliofemoral had an attempted implant procedure. A total of 1119 High Risk subjects were enrolled; however, 1108 subjects had an attempted implant procedure. The baseline data presented are for subjects with an attempted implant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk | Total
Number analyzed (Participants) | 1257 | 367 | 1108 | 2732
Age, Continuous [Mean (Standard Deviation); unit: years] — Participant Population= Consisted of all subjects with an attempted implant procedure.
  years | 83.5 (8.1) | 81.9 (8.2) | 83.6 (7.1) | 83.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Participant Population= Consisted of all subjects with an attempted implant procedure.
  Participants
    Female | 568 | 185 | 456 | 1209
    Male | 689 | 182 | 652 | 1523
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participant Population= Consisted of all subjects with an attempted implant procedure.
  Participants
    Hispanic or Latino | 37 | 4 | 38 | 79
    Not Hispanic or Latino | 1206 | 360 | 1056 | 2622
    Unknown or Not Reported | 14 | 3 | 14 | 31
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Participant Population= Consisted of all subjects with an attempted implant procedure.
  m^2 | 1.9 (0.3) | 1.8 (0.3) | 1.9 (0.2) | 1.9 (0.3)
New York Heart Association (NYHA) Classification [Number; unit: participants] — NYHA Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  participants
    NYHA Classification I | 0 | 0 | 0 | 0
    NYHA Classification II | 159 | 45 | 180 | 384
    NYHA Classification III | 881 | 248 | 811 | 1940
    NYHA Classification IV | 217 | 74 | 117 | 408
Society of Thoracic Surgeons (STS) Risk Score [Mean (Standard Deviation); unit: Percent of predicted mortality] — The Society of Thoracic Surgeons (STS) risk model predicts the risk of operative mortality and morbidity after adult cardiac surgery on the basis of patient demographic and clinical variables. After information has been entered on a given case, the online STS risk calculator provides a risk percentage for each of the outcomes. The risk percentage estimates the chance of a specific outcome for a patient with the indicated risk factors. A higher score indicates a higher risk. A lower score indicates a lower risk.
  Percent of predicted mortality | 9.1 (5.1) | 10.2 (5.6) | 7.7 (3.3) | 8.7 (4.6)
Logistic European System for Cardiac Operative Risk Evaluation (EuroSCORE) [Mean (Standard Deviation); unit: Percent of predicted mortality] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE) is a method of calculating predicted operative mortality for patients undergoing cardiac surgery. If a risk factor is present, a weight/number is assigned. The weights are added to give an approximate percent of predicted mortality. A higher score indicates a higher risk. A lower score indicates a lower risk.
  Percent of predicted mortality | 24.2 (17.1) | 24.2 (17.1) | 20.3 (13.5) | 22.6 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Extreme Risk: All-cause Death or Major Stroke; High Risk Surgical: All-cause Mortality
Description: All-cause Death or Major Stroke (Extreme Risk- Medtronic CoreValve® System); All-cause Mortality (High Risk Surgical- Medtronic CoreValve® System vs. Surgical Valve)
Time Frame: 1 year
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
percentage of participants, Kaplan-Meier | 22.5 | 30.8 | 17.8

2. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: MACCE is defined as a composite of:
  * All-Cause Death
  * Myocardial Infarction (MI)
  * All Stroke
  * Reintervention (defined as any cardiac surgery or percutaneous reintervention catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve)
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
percentage of participants, Kaplan-Meier
  30 day | 9.1 | 16.1 | 8.9
  6 month | 19.2 | 28.4 | 17.2
  1 year | 26.6 | 36.2 | 24.3

3. Secondary Outcome: The Occurrence of Individual MACCE Components
Description: Individual MACCE Components Include:
  * All Cause Mortality
  * MI
  * All stroke
  * Reintervention (defined as any cardiac surgery or percutaneous reintervention catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve)
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
percentage of participants, Kaplan-Meier
  30 day All Cause Mortality | 4.5 | 9.6 | 4.9
  30 day MI | 1.1 | 1.4 | 0.4
  30 day Stroke | 4.6 | 5.9 | 4.7
  30 day Reintervention | 0.6 | 0.8 | 0.4
  6 month All Cause Mortality | 13.7 | 20.8 | 12.0
  6 month MI | 1.6 | 2.7 | 1.0
  6 month Stroke | 6.6 | 8.2 | 7.0
  6 month Reintervention | 0.9 | 0.8 | 0.8
  1 year All Cause Mortality | 21.0 | 29.4 | 17.8
  1 year MI | 2.2 | 3.8 | 1.9
  1 year Stroke | 7.3 | 9.2 | 8.7
  1 year Reintervention | 1.0 | 1.2 | 0.8

4. Secondary Outcome: Major Adverse Events (MAEs)
Description: MAEs Include:
  * MACCE
  * Acute Kidney Injury
  * Cardiac Tamponade
  * Prosthetic Valve Dysfunction
  * Cardiogenic Shock
  * Valve Endocarditis
  * Life-Threatening, Disabling or Major Bleeding
  * Major Vascular Complication
  * Cardiac Perforation
  * Device Migration/Valve Embolism
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
percentage of participants, Kaplan-Meier
  30 day | 46.3 | 67.4 | 48.1
  6 month | 53.0 | 73.1 | 54.5
  1 year | 57.7 | 76.4 | 59.3

5. Secondary Outcome: Conduction Disturbance Requiring Permanent Pacemaker Implantation
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
percentage of participants, Kaplan-Meier
  30 day | 27.2 | 23.0 | 28.8
  6 month | 29.7 | 24.6 | 30.5
  1 year | 31.1 | 25.5 | 32.1

6. Secondary Outcome: Change From Baseline in NYHA Class
Description: Change from baseline (continuous variable). A positive number corresponds to NYHA worsening; a negative number corresponds to NYHA improvement.
  NYHA Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
Time Frame: Baseline to 30 days, baseline to 6 months, baseline to 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: average classification level change
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
average classification level change
  Baseline to 30 days | -1.2 (0.8) | -1.1 (0.9) | -1.2 (0.8)
  Baseline to 6 month | -1.4 (0.8) | -1.4 (0.8) | -1.4 (0.8)
  Baseline to 1 year | -1.4 (0.8) | -1.4 (0.9) | -1.4 (0.8)

7. Secondary Outcome: Change From Baseline in Distance Walked During 6-Minute Walk Test (6MWT)
Description: Change in distance walked during 6MWT from baseline
Time Frame: Baseline to 30 days, baseline to 1 year
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
meters
  Baseline to 30 day | 46.3 (116.4) | 4.0 (110.4) | 38.1 (100.0)
  Baseline to 1 year | 58.8 (121.2) | 28.5 (137.4) | 55.5 (117.9)

8. Secondary Outcome: Ratio of Days Alive Out of Hospital at 365 Days Post Procedure Versus Total Days Alive
Time Frame: 1 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: ratio of days alive and out of hospital
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
ratio of days alive and out of hospital | 0.8 (0.3) | 0.7 (0.4) | 0.8 (0.3)

9. Secondary Outcome: Quality of Life (QoL) Change
Description: QoL summary score change from baseline using the following measures:
  * Kansas City Cardiomyopathy Questionnaire (KCCQ): Quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
  * 12 Item Short Form Health Survey (SF-12): Measures functional health and well-being. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
  * European QoL (EQ-5D): Measures 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that can be converted to utilities using an algorithm. Utilities range from 0 to 1, with 1 representing perfect health, and 0 corresponding to the worst imaginable health state.
Time Frame: 30 day, 6 month, 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
units on a scale
  30 day KCCQ- Overall | 26.3 (26.4) | 19.9 (29.8) | 19.9 (25.0)
  30 day KCCQ- Clinical | 21.7 (26.6) | 16.5 (30.2) | 16.6 (24.0)
  30 day SF-12-Physical | 7.1 (10.7) | 5.1 (10.7) | 5.7 (10.2)
  30 day SF-12-Mental | 6.0 (13.9) | 4.5 (14.5) | 3.0 (12.4)
  30 day EQ-5D | 0.10 (0.26) | 0.07 (0.30) | 0.05 (0.21)
  6 month KCCQ- Overall | 31.7 (27.3) | 29.6 (28.5) | 26.2 (25.0)
  6 month KCCQ- Clinical | 25.8 (27.7) | 23.2 (28.5) | 20.8 (24.7)
  6 month SF-12-Physical | 7.6 (11.1) | 6.8 (11.4) | 7.1 (10.7)
  6 month SF-12-Mental | 6.9 (13.9) | 7.9 (14.9) | 4.4 (11.8)
  6 month EQ-5D | 0.10 (0.25) | 0.11 (0.27) | 0.06 (0.21)
  1 year KCCQ- Overall | 30.0 (27.5) | 28.7 (27.5) | 27.1 (24.7)
  1 year KCCQ- Clinical | 23.8 (27.9) | 21.7 (27.2) | 21.0 (24.0)
  1 year SF-12-Physical | 6.6 (11.7) | 6.4 (11.4) | 6.6 (11.1)
  1 year SF-12-Mental | 6.6 (13.9) | 6.4 (13.8) | 4.7 (12.3)
  1 year EQ-5D | 0.08 (0.26) | 0.08 (0.27) | 0.05 (0.21)

10. Secondary Outcome: Echocardiographic Assessment of Valve Performance
Description: Using the following measure:
  • Effective Orifice Area (EOA) analyzed overall per Extreme Risk or High Risk. Iliofemoral access and non-iliofemoral access are not reported separate because this is a valve performance measurement.
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with a valve implanted.
Measure: Mean (Standard Deviation); unit: cm^2
Groups:
- Extreme Risk: Implanted Cohort: Extreme Risk Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- High Risk: Implanted Cohort: High Risk Surgical Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
Arm/Group | Extreme Risk: Implanted Cohort | High Risk: Implanted Cohort
Number analyzed (Participants) | 1615 | 1102
cm^2
  30 day | 1.77 (0.53) | 1.77 (0.51)
  6 month | 1.75 (0.54) | 1.78 (0.49)
  1 year | 1.78 (0.54) | 1.77 (0.51)

11. Secondary Outcome: Echocardiographic Assessment of Valve Performance
Description: Using the following measure:
  • Transvalvular Mean Gradient analyzed overall per Extreme Risk or High Risk. Iliofemoral access and non-iliofemoral access are not reported separate because this is a valve performance measurement.
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population= Consisted of all subjects with a valve implanted.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Extreme Risk: Implanted Cohort | High Risk: Implanted Cohort
Number analyzed (Participants) | 1615 | 1102
mmHg
  30 day | 8.20 (4.26) | 8.02 (3.53)
  6 month | 7.98 (3.63) | 7.97 (3.48)
  1 year | 7.72 (3.40) | 8.12 (3.93)

12. Secondary Outcome: Echocardiographic Assessment of Valve Performance
Description: Using the following measure:
  - Degree of Aortic Valve Regurgitation (Transvalvular and Paravalvular) analyzed overall per Extreme Risk or High Risk. Iliofemoral access and non-iliofemoral access are not reported separate because this is a valve performance measurement.
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with a valve implanted.
Measure: Number; unit: percentage of participants
Arm/Group | Extreme Risk: Implanted Cohort | High Risk: Implanted Cohort
Number analyzed (Participants) | 1615 | 1102
percentage of participants
  30 day Total Aortic Regurgitation- None | 26.5 | 28.7
  30 day Total Aortic Regurgitation- Mild | 66.3 | 65.2
  30 day Total Aortic Regurgitation- Moderate | 6.9 | 5.8
  30 day Total Aortic Regurgitation- Severe | 0.3 | 0.3
  6 month Total Aortic Regurgitation- None | 35.1 | 37.8
  6 month Total Aortic Regurgitation- Mild | 58.5 | 58.1
  6 month Total Aortic Regurgitation- Moderate | 6.1 | 4.0
  6 month Total Aortic Regurgitation- Severe | 0.2 | 0.1
  1 year Total Aortic Regurgitation- None | 39.8 | 39.9
  1 year Total Aortic Regurgitation- Mild | 54.9 | 56.0
  1 year Total Aortic Regurgitation- Moderate | 5.1 | 3.8
  1 year Total Aortic Regurgitation- Severe | 0.2 | 0.3

13. Secondary Outcome: Aortic Valve Hospitalizations
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
percentage of participants, Kaplan-Meier
  30 day | 6.2 | 5.5 | 5.6
  6 month | 12.5 | 12.9 | 11.8
  1 year | 17.1 | 16.5 | 15.4

14. Secondary Outcome: Cardiovascular Deaths and Valve-Related Deaths
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
percentage of participants, Kaplan-Meier
  30 day Cardiovascular Deaths | 4.4 | 9.3 | 4.6
  30 day Valve Related Deaths | 1.9 | 4.2 | 2.4
  6 month Cardiovascular Deaths | 11.3 | 16.3 | 9.4
  6 month Valve Related Deaths | 3.9 | 5.7 | 3.8
  1 year Cardiovascular Deaths | 16.6 | 22.0 | 13.0
  1 year Valve Related Deaths | 5.5 | 6.4 | 4.2

15. Secondary Outcome: Strokes and Transient Ischemic Attacks (TIAs)
Description: Strokes (of any severity) and TIAs
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
percentage of participants, Kaplan-Meier
  30 day Stroke | 4.6 | 5.9 | 4.7
  30 day TIA | 0.7 | 0.3 | 0.7
  6 month Stroke | 6.6 | 8.2 | 6.8
  6 month TIA | 1.4 | 0.9 | 2.2
  1 year Stroke | 7.3 | 9.2 | 8.7
  1 year TIA | 2.0 | 0.9 | 2.9

16. Secondary Outcome: Index Procedure Related MAEs
Time Frame: Procedure
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
percentage of participants | 46.4 | 66.6 | 48.1

17. Secondary Outcome: Length of Index Procedure Hospital Stay
Time Frame: Number of days from admission to discharge
Population: Participant Population = Consisted of all subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1257 | 367 | 1108
days | 7.6 (6.9) | 10.7 (8.7) | 7.6 (5.9)

18. Secondary Outcome: Device Success
Description: Defined as:
  * Successful vascular access, delivery and deployment of the device, and successful retrieval of the delivery system,
  * Correct position of the device in the proper anatomical location (placement in the annulus with no impedance on device function),
  * Intended performance of the prosthetic valve (aortic valve area > 1.2 cm2 for 26, 29 and 31mm valves, ≥ 0.9 cm2 for 23mm valve (by echocardiography using the continuity equation) and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/sec, without moderate or severe prosthetic valve aortic regurgitation)
  * Only one valve implanted in the proper anatomical location
Time Frame: Number of days from admission to discharge
Population: Participant Population= Consisted of all subjects with a TAVR index procedure who were evaluable for device success.
Measure: Number; unit: percentage of participants
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1252 | 365 | 1104
percentage of participants | 84.9 | 88.1 | 87.9

19. Secondary Outcome: Procedural Success
Description: Defined as device success and absence of in-hospital MACCE.
Time Frame: Number of days from admission to discharge
Population: Participant Population = Consisted of all subjects with an index procedure who were evaluable for procedural success.
Measure: Number; unit: percentage of participants
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1252 | 365 | 1104
percentage of participants | 79.7 | 76.8 | 82.3

20. Secondary Outcome: Prosthetic Valve Dysfunction (PVD)
Description: PVD was defined according to VARC using the site reported echocardiography assessments including aortic regurgitation (AR) and aortic stenosis (AS) evaluations. Total AR reported as moderate or severe was considered PVD. AS was defined as significant stenosis and considered PVD if one of the following was met:
  * Peak velocity >4 m/s
  * Mean gradient >35 mmHg
  * EOA < 0.8 cm2
  * TVIV1 / TVIV2 < 0.25
Time Frame: 30 day, 6 months, and 1 year. The 2-5 year outcome data will be reported once data set is complete.
Population: Participant Population = Consisted of all subjects with a valve implanted.
Measure: Number; unit: Percentage of participants
Arm/Group | Extreme Risk: Iliofemoral | Extreme Risk: Non-Iliofemoral | High Risk
Number analyzed (Participants) | 1251 | 364 | 1102
Percentage of participants
  30 day Aortic Stenosis | 1.0 | 0.8 | 0.9
  30 day Aortic Regurgitation | 3.0 | 1.9 | 2.0
  6 month Aortic Stenosis | 2.2 | 0.8 | 2.0
  6 month Aortic Regurgitation | 5.0 | 3.3 | 3.1
  1 year Aortic Stenosis | 2.8 | 1.6 | 2.5
  1 year Aortic Regurgitation | 5.8 | 3.8 | 4.5

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from study enrollment to study closure, up to 5 years.
Description: All new or worsening AEs were collected through1 year. After 1 year, serious AEs, major AEs, cardiovascular events, device-related AEs, device related technical observations, unanticipated adverse device effects, strokes, and deaths were collected. AE data reported are Clinical Event Committee adjudicated AEs for subjects with an attempted implant.
Groups:
- Extreme Risk: TAVI Iliofemoral: Extreme Risk Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI); Iliofemoral Access
  Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- Extreme Risk: TAVI Non-Iliofemoral: Extreme Risk Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI); Non-Iliofemoral Access
  Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- High Risk: TAVI: High Risk Surgical Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI
Serious Adverse Events (participants affected / at risk) | 1117/1257 | 359/367 | 1004/1108
Other Adverse Events (participants affected / at risk) | 1097/1257 | 327/367 | 1001/1108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extreme Risk: TAVI Iliofemoral (N=1257) | Extreme Risk: TAVI Non-Iliofemoral (N=367) | High Risk: TAVI (N=1108)
Anaemia Deficiencies (Blood and lymphatic system disorders) | 7 (7) | 3 (3) | 6 (6)
Anaemias Due To Chronic Disorders (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 2 (2)
Anaemias (Blood and lymphatic system disorders) | 340 (420) | 150 (182) | 265 (319)
Coagulopathies (Blood and lymphatic system disorders) | 9 (9) | 6 (6) | 6 (6)
Haemolyses (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Leukocytoses (Blood and lymphatic system disorders) | 9 (9) | 4 (4) | 13 (13)
Lymphatic System Disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Marrow Depression And Hypoplastic Anaemias (Blood and lymphatic system disorders) | 3 (3) | 4 (7) | 2 (2)
Spleen Disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Thrombocytopenias (Blood and lymphatic system disorders) | 34 (34) | 17 (17) | 20 (21)
Aortic Valvular Disorders (Cardiac disorders) | 143 (153) | 26 (29) | 103 (108)
Cardiac Conduction Disorders (Cardiac disorders) | 293 (311) | 63 (66) | 277 (296)
Cardiac Disorders (Cardiac disorders) | 13 (13) | 5 (5) | 13 (13)
Cardiac Signs And Symptoms (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
Cardiac Valve Disorders (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathies (Cardiac disorders) | 16 (16) | 3 (3) | 6 (7)
Coronary Artery Disorders (Cardiac disorders) | 26 (28) | 7 (8) | 10 (11)
Heart Failures (Cardiac disorders) | 329 (531) | 105 (147) | 248 (346)
Ischaemic Coronary Artery Disorders (Cardiac disorders) | 91 (102) | 26 (30) | 78 (97)
Left Ventricular Failures (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral Valvular Disorders (Cardiac disorders) | 36 (37) | 3 (3) | 28 (30)
Myocardial Disorders (Cardiac disorders) | 6 (6) | 5 (5) | 9 (9)
Pericardial Disorders (Cardiac disorders) | 22 (24) | 8 (9) | 30 (33)
Pulmonary Valvular Disorders (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Rate And Rhythm Disorders (Cardiac disorders) | 75 (77) | 20 (21) | 50 (54)
Right Ventricular Failures (Cardiac disorders) | 4 (4) | 1 (1) | 4 (4)
Supraventricular Arrhythmias (Cardiac disorders) | 152 (184) | 47 (55) | 119 (137)
Tricuspid Valvular Disorders (Cardiac disorders) | 11 (11) | 1 (1) | 5 (5)
Ventricular Arrhythmias And Cardiac Arrest (Cardiac disorders) | 139 (150) | 43 (49) | 104 (113)
Cardiac Malpositions Congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Septal Defects Congenital (Congenital, familial and genetic disorders) | 2 (3) | 0 (0) | 3 (3)
Cardiovascular Disorders Congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Male Reproductive Tract Disorders Congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular Anomalies Congenital (Congenital, familial and genetic disorders) | 2 (2) | 1 (1) | 0 (0)
Eustachian Tube Disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
External Ear Disorders (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Inner Ear Signs And Symptoms (Ear and labyrinth disorders) | 7 (7) | 3 (3) | 2 (2)
Middle Ear Disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid Disorders (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Thyroid Hyperfunction Disorders (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Thyroid Hypofunction Disorders (Endocrine disorders) | 1 (1) | 0 (0) | 4 (4)
Blindness (Excl Colour Blindness) (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract Conditions (Eye disorders) | 5 (6) | 0 (0) | 6 (6)
Conjunctival And Corneal Bleeding And Vascular Disorders (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal Structural Change, Deposit And Degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lens Structural Change, Deposit And Degeneration (Excl Cataracts) (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lid, Lash And Lacrimal Structural Disorders (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular Bleeding And Vascular Disorders (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Partial Vision Loss (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal Bleeding And Vascular Disorders (Excl Retinopathy) (Eye disorders) | 3 (3) | 0 (0) | 4 (4)
Retinal Structural Change, Deposit And Degeneration (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
Retinal, Choroid And Vitreous Infections And Inflammations (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual Disorders (Eye disorders) | 2 (2) | 2 (2) | 3 (3)
Abdominal Findings Abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Hernias, Site Unspecified (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Abdominal Wall Conditions (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Acute And Chronic Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anal And Rectal Pains (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Benign Neoplasms Gastrointestinal (Excl Oral Cavity) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Colitis (Excl Infective) (Gastrointestinal disorders) | 4 (5) | 3 (3) | 4 (4)
Dental And Periodontal Infections And Inflammations (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dental Disorders (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diaphragmatic Hernias (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Excl Infective) (Gastrointestinal disorders) | 9 (9) | 2 (2) | 5 (5)
Diverticula (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4)
Duodenal And Small Intestinal Stenosis And Obstruction (Gastrointestinal disorders) | 7 (7) | 1 (1) | 5 (7)
Duodenal Ulcers And Perforation (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Dyspeptic Signs And Symptoms (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faecal Abnormalities (Gastrointestinal disorders) | 2 (2) | 0 (0) | 9 (9)
Flatulence, Bloating And Distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastric And Oesophageal Haemorrhages (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
Gastric Ulcers And Perforation (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0)
Gastritis (Excl Infective) (Gastrointestinal disorders) | 5 (5) | 3 (3) | 2 (2)
Gastrointestinal And Abdominal Pains (Excl Oral And Throat) (Gastrointestinal disorders) | 17 (19) | 4 (4) | 14 (15)
Gastrointestinal Atonic And Hypomotility Disorders (Gastrointestinal disorders) | 14 (15) | 0 (0) | 6 (7)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Dyskinetic Disorders (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Fistulae (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal Inflammatory Disorders (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Necrosis And Gangrene (Excl Gangrenous Hernia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal Signs And Symptoms (Gastrointestinal disorders) | 35 (35) | 12 (13) | 16 (17)
Gastrointestinal Stenosis And Obstruction (Gastrointestinal disorders) | 3 (3) | 2 (2) | 7 (7)
Gastrointestinal Ulcers And Perforation, Site Unspecified (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
Gastrointestinal Vascular Occlusion And Infarction (Gastrointestinal disorders) | 3 (3) | 2 (2) | 6 (6)
Gingival Disorders (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids And Gastrointestinal Varices (Excl Oesophageal) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Inguinal Hernias (Gastrointestinal disorders) | 5 (6) | 2 (2) | 5 (5)
Intestinal Haemorrhages (Gastrointestinal disorders) | 9 (10) | 3 (3) | 9 (9)
Intestinal Ulcers And Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2)
Large Intestinal Stenosis And Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea And Vomiting Symptoms (Gastrointestinal disorders) | 11 (11) | 6 (8) | 12 (12)
Non-Site Specific Gastrointestinal Haemorrhages (Gastrointestinal disorders) | 98 (121) | 26 (35) | 71 (84)
Oesophageal Disorders (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oesophageal Stenosis And Obstruction (Gastrointestinal disorders) | 6 (6) | 0 (0) | 1 (2)
Oesophageal Ulcers And Perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophagitis (Excl Infective) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peritoneal And Retroperitoneal Disorders (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (4)
Peritoneal And Retroperitoneal Haemorrhages (Gastrointestinal disorders) | 5 (5) | 1 (1) | 9 (9)
Tongue Disorders (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical Hernias (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Administration Site Reactions (General disorders) | 2 (2) | 0 (0) | 2 (2)
Asthenic Conditions (General disorders) | 31 (33) | 8 (10) | 23 (25)
Body Temperature Altered (General disorders) | 2 (2) | 1 (1) | 1 (1)
Complications Associated With Device (General disorders) | 5 (5) | 1 (1) | 7 (9)
Death And Sudden Death (General disorders) | 49 (49) | 18 (18) | 38 (38)
Device Issues (General disorders) | 130 (140) | 17 (19) | 93 (103)
Device Malfunction Events (General disorders) | 7 (7) | 2 (2) | 7 (7)
Device Physical Property And Chemical Issues (General disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile Disorders (General disorders) | 24 (24) | 5 (5) | 15 (15)
Gait Disturbances (General disorders) | 3 (3) | 0 (0) | 2 (2)
General Signs And Symptoms (General disorders) | 20 (20) | 4 (4) | 11 (11)
Healing Abnormal (General disorders) | 4 (4) | 1 (1) | 1 (1)
Hernias (General disorders) | 1 (1) | 0 (0) | 2 (2)
Implant And Catheter Site Reactions (General disorders) | 4 (5) | 1 (2) | 9 (9)
Inflammations (General disorders) | 2 (2) | 0 (0) | 5 (5)
Injection Site Reactions (General disorders) | 1 (1) | 0 (0) | 1 (1)
Mucosal Findings Abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 31 (32) | 7 (8) | 15 (17)
Pain And Discomfort (General disorders) | 67 (85) | 14 (18) | 40 (41)
Product Physical Issues (General disorders) | 6 (6) | 0 (0) | 0 (0)
Therapeutic And Nontherapeutic Responses (General disorders) | 1 (1) | 1 (1) | 3 (3)
Ulcers (General disorders) | 0 (0) | 0 (0) | 2 (2)
Vascular Complications Associated With Device (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bile Duct Infections And Inflammations (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis And Cholelithiasis (Hepatobiliary disorders) | 11 (11) | 4 (4) | 7 (7)
Cholestasis And Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Gallbladder Disorders (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic And Hepatobiliary Disorders (Hepatobiliary disorders) | 1 (1) | 2 (2) | 1 (1)
Hepatic Failure And Associated Disorders (Hepatobiliary disorders) | 7 (7) | 0 (0) | 5 (5)
Hepatic Fibrosis And Cirrhosis (Hepatobiliary disorders) | 4 (4) | 0 (0) | 0 (0)
Hepatic Vascular Disorders (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary Signs And Symptoms (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular Damage And Hepatitis (Hepatobiliary disorders) | 4 (4) | 1 (1) | 5 (5)
Obstructive Bile Duct Disorders (Excl Neoplasms) (Hepatobiliary disorders) | 4 (4) | 3 (3) | 1 (1)
Acute And Chronic Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic Conditions (Immune system disorders) | 1 (1) | 0 (0) | 2 (2)
Allergies To Foods, Food Additives, Drugs And Other Chemicals (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal And Gastrointestinal Infections (Infections and infestations) | 14 (14) | 2 (2) | 9 (9)
Aspergillus Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atypical Mycobacterial Infections (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bacterial Infections (Infections and infestations) | 54 (66) | 17 (22) | 37 (42)
Bone And Joint Infections (Infections and infestations) | 11 (12) | 2 (2) | 7 (7)
Candida Infections (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Cardiac Infections (Infections and infestations) | 15 (16) | 5 (5) | 10 (10)
Clostridia Infections (Infections and infestations) | 19 (23) | 9 (12) | 11 (13)
Dental And Oral Soft Tissue Infections (Infections and infestations) | 2 (2) | 1 (1) | 3 (5)
Ear Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobacter Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterococcal Infections (Infections and infestations) | 2 (2) | 1 (1) | 3 (4)
Escherichia Infections (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Eye And Eyelid Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Haemophilus Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Helicobacter Infections (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hepatobiliary And Spleen Infections (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Herpes Viral Infections (Infections and infestations) | 4 (4) | 0 (0) | 5 (5)
Infections (Infections and infestations) | 28 (30) | 8 (8) | 20 (22)
Infectious Disorders Carrier (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infectious Transmissions (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza Viral Infections (Infections and infestations) | 14 (14) | 2 (2) | 11 (12)
Klebsiella Infections (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Lower Respiratory Tract And Lung Infections (Infections and infestations) | 170 (218) | 61 (73) | 101 (116)
Male Reproductive Tract Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pseudomonal Infections (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Respiratory Syncytial Viral Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Salmonella Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis, Bacteraemia, Viraemia And Fungaemia (Infections and infestations) | 113 (133) | 35 (37) | 82 (87)
Skin Structures And Soft Tissue Infections (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Staphylococcal Infections (Infections and infestations) | 15 (17) | 4 (5) | 8 (8)
Streptococcal Infections (Infections and infestations) | 1 (1) | 2 (2) | 5 (5)
Upper Respiratory Tract Infections (Infections and infestations) | 8 (8) | 0 (0) | 7 (7)
Urinary Tract Infections (Infections and infestations) | 112 (132) | 25 (32) | 58 (67)
Vascular Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral Infections (Infections and infestations) | 6 (6) | 3 (3) | 2 (2)
Abdominal Injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Cardiac And Vascular Procedural Complications (Injury, poisoning and procedural complications) | 37 (38) | 7 (7) | 27 (27)
Cardiovascular Injuries (Injury, poisoning and procedural complications) | 9 (9) | 3 (3) | 3 (3)
Cerebral Injuries (Injury, poisoning and procedural complications) | 16 (17) | 4 (5) | 11 (13)
Chest And Lung Injuries (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2)
Ear Injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eye Injuries (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Fractures And Dislocations (Injury, poisoning and procedural complications) | 7 (8) | 0 (0) | 1 (1)
Gastrointestinal And Hepatobiliary Procedural Complications (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Limb Injuries (Incl Traumatic Amputation) (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 5 (5)
Lower Limb Fractures And Dislocations (Injury, poisoning and procedural complications) | 69 (73) | 9 (9) | 28 (28)
Muscle, Tendon And Ligament Injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Nerve Injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Neurological And Psychiatric Procedural Complications (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Non-Site Specific Injuries (Injury, poisoning and procedural complications) | 63 (67) | 16 (16) | 48 (51)
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 78 (82) | 25 (29) | 52 (54)
Overdoses (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Pelvic Fractures And Dislocations (Injury, poisoning and procedural complications) | 9 (9) | 0 (0) | 4 (4)
Poisoning And Toxicity (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 5 (5)
Renal And Urinary Tract Injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Respiratory Tract And Thoracic Cavity Procedural Complications (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Site Specific Injuries (Injury, poisoning and procedural complications) | 8 (8) | 1 (1) | 5 (5)
Skin Injuries (Injury, poisoning and procedural complications) | 21 (24) | 6 (8) | 12 (13)
Skull Fractures, Facial Bone Fractures And Dislocations (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Spinal Fractures And Dislocations (Injury, poisoning and procedural complications) | 18 (18) | 1 (1) | 7 (9)
Thermal Burns (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thoracic Cage Fractures And Dislocations (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 3 (3)
Transfusion Related Complications (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Upper Limb Fractures And Dislocations (Injury, poisoning and procedural complications) | 11 (13) | 3 (3) | 12 (14)
Urinary Tract Procedural Complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood Counts (Investigations) | 7 (7) | 0 (0) | 4 (4)
Blood Gas And Acid Base Analyses (Investigations) | 6 (6) | 7 (7) | 1 (1)
Carbohydrate Tolerance Analyses (Incl Diabetes) (Investigations) | 1 (1) | 1 (1) | 7 (7)
Cardiac Function Diagnostic Procedures (Investigations) | 16 (16) | 4 (4) | 17 (17)
Coagulation And Bleeding Analyses (Investigations) | 22 (22) | 6 (6) | 14 (17)
Ecg Investigations (Investigations) | 3 (3) | 3 (3) | 1 (1)
Faecal Analyses (Investigations) | 2 (2) | 1 (1) | 1 (1)
Heart Rate And Pulse Investigations (Investigations) | 4 (4) | 0 (0) | 2 (2)
Hepatobiliary Histopathology Procedures (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver Function Analyses (Investigations) | 2 (2) | 2 (2) | 1 (1)
Metabolism Tests (Investigations) | 0 (0) | 1 (1) | 1 (1)
Mineral And Electrolyte Analyses (Investigations) | 1 (1) | 0 (0) | 3 (4)
Musculoskeletal And Soft Tissue Histopathology Procedures (Investigations) | 1 (1) | 0 (0) | 0 (0)
Physical Examination Procedures (Investigations) | 3 (3) | 2 (2) | 0 (0)
Platelet Analyses (Investigations) | 3 (3) | 1 (1) | 0 (0)
Protein Analyses (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red Blood Cell Analyses (Investigations) | 11 (12) | 5 (5) | 8 (9)
Renal Function Analyses (Investigations) | 10 (10) | 1 (1) | 5 (5)
Respiratory And Pulmonary Function Diagnostic Procedures (Investigations) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract And Thoracic Imaging Procedures (Investigations) | 1 (1) | 0 (0) | 1 (1)
Skeletal And Cardiac Muscle Analyses (Investigations) | 9 (10) | 3 (3) | 5 (5)
Urinalysis (Investigations) | 1 (1) | 0 (0) | 2 (2)
Urinary Tract Function Analyses (Investigations) | 5 (5) | 2 (2) | 5 (5)
Vascular Auscultatory Investigations (Investigations) | 3 (3) | 0 (0) | 0 (0)
Vascular Tests (Incl Blood Pressure) (Investigations) | 8 (9) | 1 (1) | 2 (2)
White Blood Cell Analyses (Investigations) | 4 (4) | 0 (0) | 2 (2)
Appetite Disorders (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Calcium Metabolism Disorders (Metabolism and nutrition disorders) | 1 (3) | 2 (2) | 3 (3)
Chloride Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes Mellitus (Incl Subtypes) (Metabolism and nutrition disorders) | 4 (4) | 2 (3) | 4 (4)
Diabetic Complications (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Disorders Of Purine Metabolism (Metabolism and nutrition disorders) | 6 (7) | 0 (0) | 8 (9)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 12 (12) | 3 (3) | 4 (4)
General Nutritional Disorders (Metabolism and nutrition disorders) | 31 (32) | 12 (12) | 10 (10)
Hyperglycaemic Conditions (Metabolism and nutrition disorders) | 18 (20) | 8 (8) | 15 (15)
Hypoglycaemic Conditions (Metabolism and nutrition disorders) | 13 (13) | 9 (10) | 8 (8)
Magnesium Metabolism Disorders (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2)
Metabolic Acidoses (Excl Diabetic Acidoses) (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 4 (4)
Metabolic Alkaloses (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Mixed Acid-Base Disorders (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Phosphorus Metabolism Disorders (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Potassium Imbalance (Metabolism and nutrition disorders) | 34 (37) | 10 (12) | 25 (26)
Protein Metabolism Disorders (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Sodium Imbalance (Metabolism and nutrition disorders) | 21 (23) | 2 (2) | 20 (23)
Total Fluid Volume Decreased (Metabolism and nutrition disorders) | 37 (37) | 13 (14) | 29 (30)
Total Fluid Volume Increased (Metabolism and nutrition disorders) | 35 (36) | 10 (10) | 23 (23)
Arthropathies (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Bone Disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Bursal Disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Connective Tissue Disorders (Excl Le) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Crystal Arthropathic Disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Extremity Deformities (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint Related Disorders (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Joint Related Signs And Symptoms (Musculoskeletal and connective tissue disorders) | 10 (10) | 3 (3) | 9 (9)
Muscle Infections And Inflammations (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Related Signs And Symptoms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Weakness Conditions (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4) | 5 (5)
Musculoskeletal And Connective Tissue Pain And Discomfort (Musculoskeletal and connective tissue disorders) | 38 (43) | 8 (8) | 23 (25)
Musculoskeletal And Connective Tissue Signs And Symptoms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Myopathies (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (3)
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 6 (8) | 1 (1) | 13 (15)
Rheumatoid Arthropathies (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Soft Tissue Disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Spine And Neck Deformities (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Tendon Disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
B-Cell Lymphomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bile Duct Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1) | 1 (1)
Bone Neoplasms Malignant (Excl Sarcomas) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast And Nipple Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 2 (2)
Burkitt's Lymphomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cardiovascular Neoplasms Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Central Nervous System Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Colonic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0) | 4 (4)
Hepatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Leiomyosarcomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Leukaemias Acute Myeloid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Leukaemias Chronic Lymphocytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Leukaemias (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Lip And Oral Cavity Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Lymphomas Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mantle Cell Lymphomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases To Specified Sites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Multiple Myelomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic Syndromes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 4 (4)
Myeloproliferative Disorders (Excl Leukaemias) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasms Malignant Site Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 3 (3) | 6 (6)
Nervous System Neoplasms Unspecified Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Non-Small Cell Neoplasms Malignant Of The Respiratory Tract Cell Type Specified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Oesophageal Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Oncologic Complications And Emergencies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic Neoplasms Malignant (Excl Islet Cell And Carcinoid) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 3 (3)
Prostatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 2 (2)
Rectal Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Renal Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
Respiratory Tract And Pleural Neoplasms Malignant Cell Type Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 7 (7) | 2 (2)
Skin Melanomas (Excl Ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Skin Neoplasms Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Skin Neoplasms Malignant And Unspecified (Excl Melanoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0) | 3 (3)
Small Intestinal Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Soft Tissue Sarcomas Histology Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine Neoplasms Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Vulval Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Acute Polyneuropathies (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Alzheimer's Disease (Incl Subtypes) (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Autonomic Nervous System Disorders (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Central Nervous System Aneurysms (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Central Nervous System Haemorrhages And Cerebrovascular Accidents (Nervous system disorders) | 98 (105) | 30 (33) | 79 (86)
Central Nervous System Vascular Disorders (Nervous system disorders) | 10 (11) | 2 (3) | 7 (7)
Cerebellar Coordination And Balance Disturbances (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Coma States (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cortical Dysfunction (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dementia (Excl Alzheimer's Type) (Nervous system disorders) | 5 (5) | 0 (0) | 5 (5)
Disturbances In Consciousness (Nervous system disorders) | 42 (46) | 13 (14) | 32 (33)
Dyskinesias And Movement Disorders (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathies (Nervous system disorders) | 27 (29) | 8 (8) | 13 (13)
Encephalopathies Toxic And Metabolic (Nervous system disorders) | 22 (22) | 1 (1) | 14 (14)
Facial Cranial Nerve Disorders (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Generalised Tonic-Clonic Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headaches (Nervous system disorders) | 10 (10) | 1 (1) | 8 (9)
Hydrocephalic Conditions (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Lumbar Spinal Cord And Nerve Root Disorders (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Memory Loss (Excl Dementia) (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Mental Impairment (Excl Dementia And Memory Loss) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mononeuropathies (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Motor Neurone Diseases (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple Sclerosis Acute And Progressive (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myelitis (Incl Infective) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurological Signs And Symptoms (Nervous system disorders) | 32 (34) | 6 (6) | 18 (19)
Neuromuscular Junction Dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paralysis And Paresis (Excl Cranial Nerve) (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
Parkinson's Disease And Parkinsonism (Nervous system disorders) | 3 (4) | 0 (0) | 1 (1)
Peripheral Neuropathies (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Seizures And Seizure Disorders (Nervous system disorders) | 12 (18) | 3 (3) | 5 (5)
Sensory Abnormalities (Nervous system disorders) | 3 (3) | 0 (0) | 5 (5)
Speech And Language Abnormalities (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal Cord And Nerve Root Disorders (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Structural Brain Disorders (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Transient Cerebrovascular Events (Nervous system disorders) | 30 (34) | 5 (6) | 24 (27)
Tremor (Excl Congenital) (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Trigeminal Disorders (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vagus Nerve Disorders (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Abnormal Behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety Disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety Symptoms (Psychiatric disorders) | 8 (10) | 4 (4) | 10 (11)
Behaviour And Socialisation Disturbances (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar Disorders (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion And Disorientation (Psychiatric disorders) | 24 (24) | 10 (10) | 20 (20)
Deliria (Psychiatric disorders) | 14 (14) | 1 (1) | 9 (9)
Delusional Symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depressive Disorders (Psychiatric disorders) | 6 (6) | 1 (1) | 4 (4)
Disturbances In Initiating And Maintaining Sleep (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Eating Disorders (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Mental Disorders (Psychiatric disorders) | 56 (64) | 19 (21) | 29 (29)
Panic Attacks And Disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Perception Disturbances (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Psychiatric Symptoms (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Speech Articulation And Rhythm Disturbances (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Stress Disorders (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Substance-Related Disorders (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal And Self-Injurious Behaviour (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1)
Bladder And Urethral Symptoms (Renal and urinary disorders) | 51 (57) | 6 (8) | 48 (49)
Bladder Disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
Genital And Urinary Tract Disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Myoneurogenic Bladder Disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Nephropathies And Tubular Disorders (Renal and urinary disorders) | 3 (3) | 0 (0) | 2 (2)
Renal Disorders (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal Failure And Impairment (Renal and urinary disorders) | 208 (263) | 76 (94) | 154 (181)
Renal Failure Complications (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Renal Lithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 6 (7)
Renal Neoplasms (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Obstructive Disorders (Renal and urinary disorders) | 4 (4) | 1 (1) | 0 (0)
Renal Vascular And Ischaemic Conditions (Renal and urinary disorders) | 2 (2) | 1 (1) | 4 (4)
Structural And Obstructive Urethral Disorders (Excl Congenital) (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3)
Ureteric Disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Abnormalities (Renal and urinary disorders) | 29 (33) | 9 (9) | 29 (36)
Urinary Tract Lithiasis (Excl Renal) (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Breast Disorders (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
Cervix Disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian And Fallopian Tube Cysts And Neoplasms (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvis And Broad Ligament Disorders (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Penile And Scrotal Infections And Inflammations (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile Disorders (Excl Erection And Ejaculation) (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Prostatic Neoplasms And Hypertrophy (Reproductive system and breast disorders) | 4 (4) | 1 (1) | 2 (2)
Prostatic Signs, Symptoms And Disorders (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Reproductive Tract Signs And Symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Scrotal Disorders (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 1 (1)
Testicular And Epididymal Disorders (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal Disorders (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal Signs And Symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Breathing Abnormalities (Respiratory, thoracic and mediastinal disorders) | 101 (121) | 31 (39) | 66 (76)
Bronchial Conditions (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (2)
Bronchospasm And Obstruction (Respiratory, thoracic and mediastinal disorders) | 55 (94) | 26 (40) | 35 (42)
Conditions Associated With Abnormal Gas Exchange (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 11 (12) | 22 (23)
Coughing And Associated Symptoms (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 6 (7) | 6 (6)
Diaphragmatic Disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal And Adjacent Sites Disorders (Excl Infections And Neoplasms) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Laryngeal Spasm, Oedema And Obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Lower Respiratory Tract Inflammatory And Immunologic Conditions (Respiratory, thoracic and mediastinal disorders) | 34 (37) | 6 (7) | 14 (15)
Lower Respiratory Tract Signs And Symptoms (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1)
Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 1 (1)
Nasal Disorders (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 11 (12) | 14 (15)
Parenchymal Lung Disorders (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 4 (4) | 10 (10)
Pharyngeal Disorders (Excl Infections And Neoplasms) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Pleural Conditions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax And Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 106 (137) | 70 (91) | 75 (92)
Pulmonary Hypertensions (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 8 (9)
Pulmonary Oedemas (Respiratory, thoracic and mediastinal disorders) | 31 (34) | 17 (17) | 35 (40)
Pulmonary Thrombotic And Embolic Conditions (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (5) | 11 (11)
Respiratory Failures (Excl Neonatal) (Respiratory, thoracic and mediastinal disorders) | 149 (192) | 66 (77) | 108 (126)
Respiratory Tract Disorders (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 1 (1)
Upper Respiratory Tract Signs And Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Bullous Conditions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermal And Epidermal Conditions (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2) | 2 (2)
Dermatitis And Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Erythemas (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Exfoliative Conditions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkeratoses (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail And Nail Bed Conditions (Excl Infections And Infestations) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Purpura And Related Conditions (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Rashes, Eruptions And Exanthems (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Skin And Subcutaneous Conditions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin And Subcutaneous Tissue Ulcerations (Skin and subcutaneous tissue disorders) | 9 (10) | 2 (2) | 7 (7)
Skin Injuries And Mechanical Dermatoses (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 1 (1)
Skin Preneoplastic Conditions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin Vasculitides (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Vasomotor Conditions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial Therapeutic Procedures (Excl Aortic) (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardiac Device Therapeutic Procedures (Surgical and medical procedures) | 8 (8) | 2 (2) | 3 (3)
Haematological Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Joint Therapeutic Procedures (Surgical and medical procedures) | 5 (5) | 1 (1) | 1 (1)
Large Intestine Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Lens Therapeutic Procedures (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Prostatic Therapeutic Procedures (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Renal Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Therapeutic Bladder Catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Therapeutic Procedures (Surgical and medical procedures) | 20 (22) | 1 (1) | 11 (11)
Tracheal Therapeutic Procedures (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Venous Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Accelerated And Malignant Hypertension (Vascular disorders) | 13 (13) | 2 (2) | 13 (13)
Aneurysms And Dissections Non-Site Specific (Vascular disorders) | 5 (5) | 2 (2) | 6 (6)
Aortic Aneurysms And Dissections (Vascular disorders) | 8 (9) | 6 (6) | 5 (5)
Aortic Embolism And Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic Necrosis And Vascular Insufficiency (Vascular disorders) | 3 (3) | 1 (1) | 1 (1)
Arterial And Aortic Injuries (Vascular disorders) | 11 (11) | 0 (0) | 10 (11)
Arterial Inflammations (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Disorders (Vascular disorders) | 4 (4) | 1 (1) | 3 (3)
Circulatory Collapse And Shock (Vascular disorders) | 7 (7) | 4 (4) | 4 (4)
Haemorrhages (Vascular disorders) | 43 (43) | 16 (16) | 33 (34)
Lymphangiopathies (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Lymphoedemas (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Non-Site Specific Embolism And Thrombosis (Vascular disorders) | 9 (10) | 4 (4) | 7 (7)
Non-Site Specific Necrosis And Vascular Insufficiency (Vascular disorders) | 6 (6) | 1 (1) | 4 (5)
Non-Site Specific Vascular Disorders (Vascular disorders) | 16 (16) | 10 (10) | 12 (12)
Peripheral Aneurysms And Dissections (Vascular disorders) | 24 (24) | 2 (2) | 11 (11)
Peripheral Embolism And Thrombosis (Vascular disorders) | 20 (20) | 8 (8) | 17 (19)
Peripheral Vascular Disorders (Vascular disorders) | 5 (6) | 5 (8) | 6 (6)
Peripheral Vasoconstriction, Necrosis And Vascular Insufficiency (Vascular disorders) | 35 (37) | 16 (17) | 41 (44)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Site Specific Necrosis And Vascular Insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Site Specific Vascular Disorders (Vascular disorders) | 3 (3) | 1 (1) | 1 (2)
Vascular Hypertensive Disorders (Vascular disorders) | 54 (60) | 22 (23) | 53 (57)
Vascular Hypotensive Disorders (Vascular disorders) | 137 (157) | 50 (52) | 90 (93)
Vascular Malformations And Acquired Anomalies (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extreme Risk: TAVI Iliofemoral (N=1257) | Extreme Risk: TAVI Non-Iliofemoral (N=367) | High Risk: TAVI (N=1108)
Anaemias (Blood and lymphatic system disorders) | 244 (259) | 92 (96) | 260 (267)
Leukocytoses (Blood and lymphatic system disorders) | 82 (88) | 38 (40) | 79 (81)
Thrombocytopenias (Blood and lymphatic system disorders) | 175 (182) | 70 (74) | 217 (223)
Cardiac Conduction Disorders (Cardiac disorders) | 286 (335) | 56 (65) | 331 (387)
Heart Failures (Cardiac disorders) | 96 (107) | 30 (31) | 68 (74)
Rate And Rhythm Disorders (Cardiac disorders) | 85 (92) | 28 (30) | 99 (105)
Supraventricular Arrhythmias (Cardiac disorders) | 153 (174) | 72 (81) | 159 (186)
Ventricular Arrhythmias And Cardiac Arrest (Cardiac disorders) | 64 (69) | 15 (16) | 66 (69)
Gastrointestinal Atonic And Hypomotility Disorders (Gastrointestinal disorders) | 66 (70) | 27 (27) | 74 (78)
Nausea And Vomiting Symptoms (Gastrointestinal disorders) | 57 (61) | 19 (22) | 45 (51)
Asthenic Conditions (General disorders) | 57 (63) | 23 (25) | 43 (44)
Febrile Disorders (General disorders) | 75 (77) | 24 (25) | 69 (71)
Oedema (General disorders) | 93 (102) | 17 (17) | 85 (95)
Pain And Discomfort (General disorders) | 72 (86) | 22 (29) | 71 (84)
Lower Respiratory Tract And Lung Infections (Infections and infestations) | 67 (75) | 22 (22) | 55 (58)
Urinary Tract Infections (Infections and infestations) | 149 (182) | 45 (46) | 141 (164)
Non-Site Specific Injuries (Injury, poisoning and procedural complications) | 86 (93) | 16 (19) | 68 (77)
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 74 (80) | 25 (27) | 87 (92)
Skeletal And Cardiac Muscle Analyses (Investigations) | 52 (54) | 25 (26) | 42 (43)
Hyperglycaemic Conditions (Metabolism and nutrition disorders) | 33 (34) | 27 (27) | 46 (46)
Magnesium Metabolism Disorders (Metabolism and nutrition disorders) | 25 (25) | 12 (14) | 64 (65)
Potassium Imbalance (Metabolism and nutrition disorders) | 84 (96) | 34 (35) | 87 (99)
Sodium Imbalance (Metabolism and nutrition disorders) | 61 (68) | 28 (29) | 58 (63)
Total Fluid Volume Increased (Metabolism and nutrition disorders) | 85 (89) | 28 (28) | 116 (122)
Musculoskeletal And Connective Tissue Pain And Discomfort (Musculoskeletal and connective tissue disorders) | 89 (100) | 29 (33) | 99 (108)
Confusion And Disorientation (Psychiatric disorders) | 57 (59) | 24 (24) | 68 (69)
Bladder And Urethral Symptoms (Renal and urinary disorders) | 35 (35) | 13 (13) | 57 (60)
Renal Failure And Impairment (Renal and urinary disorders) | 165 (199) | 58 (66) | 201 (223)
Breathing Abnormalities (Respiratory, thoracic and mediastinal disorders) | 77 (81) | 16 (18) | 64 (67)
Parenchymal Lung Disorders (Respiratory, thoracic and mediastinal disorders) | 72 (75) | 25 (25) | 94 (98)
Pneumothorax And Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 138 (146) | 64 (73) | 168 (187)
Pulmonary Oedemas (Respiratory, thoracic and mediastinal disorders) | 68 (70) | 14 (14) | 67 (69)
Haemorrhages (Vascular disorders) | 55 (57) | 9 (9) | 61 (62)
Vascular Hypertensive Disorders (Vascular disorders) | 146 (152) | 56 (58) | 192 (206)
Vascular Hypotensive Disorders (Vascular disorders) | 146 (162) | 45 (49) | 120 (131)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less